CLINICAL TRIAL: NCT01203332
Title: Identifying Undiagnosed Asymptomatic HIV Infection in Hispanic/Latino Adolescents and Young Adults
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 096
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HIV
Keywords: HIV testing; Latino; Latina; Men who have sex with men
MeSH Terms: conditions — Homosexuality | interventions — HIV Testing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Alternative Venue Testing (AVT): Participants recruited for testing through the AVT recruitment method.
  Interventions: Behavioral: Effectiveness of different strategies in HIV testing and linkage to care
- SSNIT - Index Recruiter: Participants recruited for HIV testing and to bring members of their social and sexual network to the study.
  Interventions: Behavioral: Effectiveness of different strategies in HIV testing and linkage to care
- SSNIT - Network Member: Participants recruited by someone in their social or sexual network to participate in the study, including HIV testing.
  Interventions: Behavioral: Effectiveness of different strategies in HIV testing and linkage to care

INTERVENTIONS:
Behavioral: Effectiveness of different strategies in HIV testing and linkage to care — HIV testing Linkage to Care

SUMMARY:
The proposed research will include adolescent and young adult Hispanic/Latino men who have sex with men (MSM) and heterosexual men and women, aged 13-24 years, and will be based at 13 ATN Adolescent Medicine Trial Units (AMTUs) that provide clinical care and psychosocial services to the target group. In 10 of the 13 sites, comparisons will be made between alternative venue-based testing (AVT) and social and sexual network-based interviewing and HIV testing (SSNIT) strategies to assess which, among these approaches, is the most effective means for identifying undiagnosed human immunodeficiency virus (HIV) in young, at-risk Hispanics/Latinos. Three of the sites will focus solely on use of SSNIT for identifying undiagnosed HIV in our target group of adolescents and young adults. All study participants will complete an audio computer-assisted self-interview (ACASI) and undergo HIV screening. Participants with presumptive HIV positive screening results will be referred to the local AMTU for confirmatory testing, post-test counseling and referrals for linkage to HIV medical care. Linkage to care for ATN 096 study participants will be conducted in accordance with the Strategic Multisite Initiative for the Identification, Linkage, and Engagement in Care of Youth with Undiagnosed HIV Infection (SMILE in CARING for YOUTH) Program (ATN 093), a collaboration of the CDC and NICHD/ATN, to ensure that youth who test positive for HIV as part of this protocol are linked with treatment and care.

ELIGIBILITY:
1. Inclusion Criteria

1a. Alternative Venue-Based Testing (AVT) Participants

* Self-identifies as being of Hispanic or Latino ethnicity;
* Provides verbal confirmation that his/her age is between 13 years, 0 days to 24 years, 364 days at the time of enrollment;
* Self-reports a negative or unknown HIV status;
* Is male and self-reports any unprotected anal sex with a male sexual partner in the past three months; OR Is female and self-reports any unprotected anal or vaginal sex with two or more male sexual partners in the past three months; OR Is female and self-reports any unprotected anal or vaginal sex with a male sexual partner who was incarcerated in the past 12 months; OR Is male or female and self-reports any history of injection drug use; OR Is male or female and self-reports any unprotected anal or vaginal sex with an individual who is known to be HIV positive; OR Is male or female and self-reports any unprotected anal or vaginal sex with an injection drug user in the past 12 months;
* Willing to complete an HIV risk assessment;
* Willing to undergo HIV screening; and
* Able to understand and willing to provide signed informed consent/assent in English or Spanish.

  1b. Social and Sexual Index Recruiter Participants
* Self-identifies as being of Hispanic or Latino ethnicity;
* Provides verbal confirmation that his/her age is between 13 years, 0 days to 24 years, 364 days at the time of enrollment;
* Is male or female and self-reports being diagnosed with HIV in the past 12 months; OR Is female and self-reports any unprotected anal or vaginal sex with a male sexual partner who was incarcerated in the past 12 months; OR Is male or female and self-reports any history of injection drug use; OR Is male or female and self-reports any unprotected anal or vaginal sex with an individual who is known to be HIV positive; OR Is male or female and self-reports any unprotected anal or vaginal sex with an injection drug user in the past 12 months;
* Willing to complete a HIV risk assessment;
* Willing to undergo HIV screening (or an HIV confirmatory test if previously diagnosed);
* Willing to recruit one or more Latino/Latina family members, friends, or sexual partners who are between the ages of 13-24 years and who meet the criteria for a Social and Sexual Network Member for participation in the study; and
* Able to understand and willing to provide signed informed consent/assent in English or Spanish.

  1c. Social and Sexual Network Members
* Self-identifies as being of Hispanic or Latino ethnicity;
* Provides verbal confirmation that his/her age is between 13 years, 0 days to 24 years, 364 days at the time of enrollment;
* Self-reports any anal or vaginal sexual activity in the past 3 months and any unprotected anal or vaginal sex in the last 12 months; OR Self-reports any history of injection drug use;
* Willing to complete a HIV risk assessment;
* Willing to undergo HIV screening; and
* Able to understand and willing to provide signed informed consent/assent in English or Spanish.

  1d. Additional Inclusion Criteria for Social and Sexual Network Member Recruiters
* Is male or female and self-reports being diagnosed with HIV in the past 12 months; OR Is female and self-reports any unprotected anal or vaginal sex with a male sexual partner who was incarcerated in the past 12 months; OR Is male or female and self-reports any history of injection drug use; OR Is male or female and self-reports any unprotected anal or vaginal sex with an individual who is known to be HIV positive; OR Is male or female and self-reports any unprotected anal or vaginal sex with an IDU in the past 12 months; and
* Willing to recruit one or more Latino/Latina family members, friends, or sexual partners who are between the ages of 13-24 years and who meet the criteria for Social and Sexual Network Members for participation in the study.

  2. Exclusion Criteria

  2a. All Participants
* Previous participation in ATN 096 as an AVT or a SSNIT study participant;
* Current or prior participation in ATN 084;
* Anything that would impair the participant's ability to provide informed consent/assent and/or interfere with the protocol's objectives; i.e., readily apparent psychiatric symptoms (hallucinations, thought disorder), visibly distraught (suicidal, homicidal, exhibiting violent behavior) or visibly intoxicated or under the influence of alcohol or other substances at the time of study enrollment, and
* Acute illness that, in the opinion of study staff, would interfere with the participant's ability to adhere to the protocol requirements and/or interfere with the protocol objectives.

  2b. Additional Exclusion Criteria for Alternative Venue-Based Testing Participants
* Self-reports a prior diagnosis of HIV

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent and young adult Hispanic/Latino MSM and heterosexual men and women, aged 13-24 years, who meet all eligibility requirements for enrollment into the AVT or SSNIT component of the study.
Sampling Method: Non-Probability Sample
Enrollment: 1917 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of AVT strategy with SSNIT | 2 years
  To compare the relative effectiveness of AVT with SSNIT, which is a coupon-based index recruiter driven network recruitment strategy for identifying previously undiagnosed HIV infection among Hispanic/Latino adolescents and young adults aged 13-24 years.
Facilitators & barriers to HIV testing | 2 years
  To examine factors that facilitate and/or hinder Hispanic/Latino adolescents and young adults in getting an HIV test (e.g., perceived risk for HIV, acculturation, homophobia, stigma associated with IDU).
Sub-group differences | 2 years
  To explore the extent to which sub-group differences (e.g., origin of birth, age, level of acculturation) exist by prevalence of HIV-related risk behaviors, HIV testing, and mode of HIV transmission.

CONTACTS AND LOCATIONS:
Overall Officials: Cherrie B. Boyer, Ph.D., Study Chair — Adolescent Trials Network; Jonathan M. Ellen, M.D., Study Chair — Adolescent Trials Network
Locations (13):
- United States (12):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Childrens Diagnostic & Treatment Center, Fort Lauderdale, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Ruth M Rothstein CORE Center/ John H Stroger Jr Hospital, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- See also: Related Info — http://www.atnonline.org